CLINICAL TRIAL: NCT04564495
Title: Home Based Tele-exercise for People With Chronic Neurological Impairments
Acronym: Telex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telex
Record Dates: First submitted 2020-09-23; First posted 2020-09-25 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Neurologic Disorder; Stroke; Spinal Cord Injuries; Cerebral Palsy; Hemiplegia; Hemiparesis; Multiple Sclerosis; Parkinson Disease; Trauma, Brain; Transverse Myelitis; Friedreich Ataxia
MeSH Terms: conditions — Nervous System Diseases; Stroke; Spinal Cord Injuries; Cerebral Palsy; Hemiplegia; Paresis; Multiple Sclerosis; Parkinson Disease; Brain Injuries, Traumatic; Myelitis, Transverse; Friedreich Ataxia

STUDY DESIGN:
Intervention Model Description: One group will attend live zoom classes with instructor feedback, and the other group will exercise using pre-recorded sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live zoom exercise classes (Experimental): Participants will engage in a live zoom exercise session. Participants will undergo 45 minutes of aerobic exercise intervention, three times a week, for a period of 12 weeks. Exercise will include repetitive bouts of high intensity exercises with intermittent periods of rest or active recovery. circuit of moves like 'jabs', 'hooks' etc, and a strength and endurance class that promotes postural awareness.
  Interventions: Behavioral: Seated exercise
- Recorded zoom exercise classes (Active Comparator): Participants will undergo 45 minutes of aerobic exercise intervention, three times a week, for a period of 12 weeks, using a pre-recorded class that they can do according to their own schedule. Exercise will include repetitive bouts of high intensity exercises with intermittent periods of rest or active recovery. circuit of moves like 'jabs', 'hooks' etc, and a strength and endurance class that promotes postural awareness.
  Interventions: Behavioral: Seated exercise

INTERVENTIONS:
Behavioral: Seated exercise — Exercise will include repetitive bouts of high intensity exercises with intermittent periods of rest or active recovery. circuit of moves like 'jabs', 'hooks' etc, and a strength and endurance class that promotes postural awareness.

SUMMARY:
To assess the impact of a 12-week virtual seated physical intervention on cardiovascular health and wellness in people with chronic neurological impairments (CNI).

DETAILED DESCRIPTION:
This study aims to examine how effective seated Zoom exercise classes are for a person with CNI for addressing cardiovascular health, physical wellness and quality of life. If these classes prove to be effective, online platforms could be a viable avenue for those with CNI to exercise and increase/maintain wellness without having to leave their homes. The investigators are also attempting to determine if a class with a live instructor vs a pre-recorded class has an effect on motivation, compliance, exertion and modifications/safety.

The entire process, including screening and consenting, will be done via Zoom and Redcap, potentially providing a blueprint for the future studies. This process can enable participants to participate in studies with minimal inconvenience, expense and effort of traveling for the consent process.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with chronic (>6 months) neurological impairments
2. 18 to 75 years of age
3. Participants who can provide a medical clearance to participate in the program
4. Participants who can remain seated for at least one hour
5. Heart rate/BP considerations, per each participant's MD
6. Participants must be able to don/doff HR monitor without assistance, or have assistance if necessary
7. Participants must maintain their current exercise/physical activity routine during the course of the study
8. Clinically stable with no other neurological, medical or cognitive impairments
9. Reliable Internet connection and ability to use Zoom platform
10. Participants must speak and understand English
11. No contraindication/limitations to exercise
12. Currently exercising 2 days or less per week

Exclusion Criteria:

1. Participants with any cognitive impairment preventing safe and accurate participation in the program
2. Medical issues preventing safe participation
3. Other problems possibly contraindicating autonomous exercise at home if no supervision available.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | Within one week before the first intervention session to within one week after the end of intervention
  Heart rate on last day of training compared to heart rate on first day of training

SECONDARY OUTCOMES:
Perceived Wellness Survey | Within one week before the first intervention session to within one week after the end of intervention
  a 36-item instrument used to measure an individual's perceived health status in physical, psychological, emotional, intellectual, spiritual, and social wellness constructs
Physical Activity Enjoyment Scale | Within one week before the first intervention session to within one week after the end of intervention
  a self-assessment measure of enjoyment with their current physical activity
Short Form-36 Health Survey | Within one week before the first intervention session to within one week after the end of intervention
  measures physical health and mental health
Numerical pain rating | Within one week before the first intervention session to within one week after the end of intervention
  standardized instrument for pain assessment in clinical and research practice. It is an 11-point scale from 0 (no pain) to 10 (the most intense pain) at rest and during movement
Borg's Rating Scale of Perceived Exertion | Within one week before the first intervention session to within one week after the end of intervention
  standardized measure to evaluate perceived intensity of exertion, effort, and fatigue during physical exercise
Reason for exercise inventory | Within one week before the first intervention session to within one week after the end of intervention
  is a 24-item scale to assess the reason that motivates a person to exercise

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Friel, Principal Investigator — Burke Medical Research Institute
Locations (1):
- Burke Neurological Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to use the concept, methods and analysis as a framework to develop evidence-based protocols for future cohorts and studies. We have made a commitment to publish all relevant scientific information in a timely manner. Unpublished information may be available to interested individuals or organizations by request to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: These types of supporting information will be published as a protocol paper, and will remain accessible with no end date.

REFERENCES:
- [Derived] Kumar DS, Bialek A, Divecha AA, Garn RM, Currie LEJ, Friel KM. A seated virtual exercise program to improve cardiovascular function in adults with chronic neurological impairments: a randomized controlled trial. Front Rehabil Sci. 2025 Mar 26;6:1477969. doi: 10.3389/fresc.2025.1477969. eCollection 2025. PMID 40207026
- [Derived] Divecha AA, Bialek A, Kumar DS, Garn RM, Currie LEJ, Campos T, Friel KM. Effects of a 12-week, seated, virtual, home-based tele-exercise programme compared with a prerecorded video-based exercise programme in people with chronic neurological impairments: protocol for a randomised controlled trial. BMJ Open. 2023 Jan 24;13(1):e065032. doi: 10.1136/bmjopen-2022-065032. PMID 36693691